CLINICAL TRIAL: NCT04227106
Title: VIITAL: A Phase 3 Study of EB-101 for the Treatment of Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Brief Title: Phase 3, Open-label Clinical Trial of EB-101 for the Treatment of Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abeona Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EB-101-CL-301
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-04

CONDITIONS: Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa
Keywords: chronic wounds
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EB-101 (Experimental): One-time surgical application of EB-101 on up to 6 chronic, RDEB wounds
  Interventions: Biological: EB-101

INTERVENTIONS:
Biological: EB-101 — autologous RDEB keratinocytes isolated from skin biopsies and transduced with a recombinant retrovirus containing a full-length COL7A1 expression cassette for C7
  Other Names: LZRSE-Col7A1 Engineered Autologous Epidermal Sheets [LEAES]

SUMMARY:
The purpose of this trial is to evaluate safety and efficacy of surgical application of EB-101 (autologous, gene-corrected keratinocyte sheets) as a treatment of recessive dystrophic epidermolysis bullosa (RDEB).

DETAILED DESCRIPTION:
Recessive dystrophic epidermolysis bullosa (RDEB) is an ultra-rare, severe inherited blistering skin disease caused by the absence of a protein known as type 7 collagen (C7). There is no approved treatment for RDEB. Only supportive care is currently possible.

This open-label, controlled study will evaluate the efficacy and safety of EB-101 for the treatment of large, chronic, RDEB wounds. The study intervention consists of one-time surgical application of gene-corrected keratinocyte sheets (EB-101) for the treatment of RDEB wound sites in up to approximately 10-15 participants. A single EB-101 sheet is able to provide healing to a wound area up to approximately 40cm2. Up to 6 (six) EB-101 sheets may be applied to each patient, depending on the area of existing wounds. The co-primary endpoints of the study are: 1) the proportion of RDEB wound sites with greater than or equal to 50% healing from baseline, comparing treated with untreated wound sites at Week 24 (Month 6) as determined by direct investigator assessment; and 2) pain reduction associated with wound dressing change assessed by the mean differences in scores of the Wong-Baker FACES scale between treated and untreated wounds at Week 24 (Month 6). Patient-reported outcomes and safety will also be collected throughout the study.

The primary analysis for efficacy will be assessed when all patients reach Week 24. Safety and efficacy assessments will be conducted at regular intervals and completed when last patient reaches Week 26 post-treatment.

Upon completion of the study period, patients will be monitored annually as per standard of care for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RDEB;
* Age 6 years or older, willing and able to give consent/assent;
* If under the age of 18, guardian(s) is/are willing and able to give consent;
* Positive expression of the non-collagenous region 1 of the type 7 collagen protein (NC1+) in the skin;
* Two confirmed RDEB C7 mutations with recessive inheritance patterns (or confirmation that parents don't have any evidence of dominant disease);
* At least 40 cm2 areas of chronically wounded area on the trunk and/or extremities suitable for EB-101 application (open erosions);
* Able to undergo adequate anesthesia during EB-101 application;
* Must have at least two matched, eligible wound sites (one pair);

  * Wound sites must:

    * Have an area ≥20 cm2,
    * Present for ≥6 months, and
    * Stage 2 wound;
* Women of childbearing potential must use a reliable birth control method throughout the duration of the study and for 6 months post treatment;
* Negative pregnancy test;
* Must be on stable pain medication regimen at least 30 days prior to Screening

Exclusion Criteria:

* Medical instability limiting ability to travel to the study site;
* The presence of medical illness expected to complicate participation and/or compromise the safety of this technique, such as active infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C;
* Evidence of immune response to C7 by indirect immunofluorescence (IIF);
* Evidence of systemic infection;
* Current evidence or a history of squamous cell carcinoma (SCC) in the area that will undergo EB-101 application;
* Active drug or alcohol addiction;
* Hypersensitivity to vancomycin or amikacin;
* Receipt of chemical or biological study product for the specific treatment of RDEB in the past 3 months;
* Positive pregnancy test or breast-feeding;
* Clinically significant medical or laboratory abnormalities as determined by the Principal Investigator;
* Inability to properly follow protocol and protect keratinocyte sheet sites, as determined by the Principal Investigator;
* Grade 3 clinical event or laboratory abnormality at Day 0. Abnormalities such as esophageal strictures, anemia, low albumin, and pain/itch are expected in RDEB patients. These abnormalities will not exclude a participant; and
* Inability to culture participant's keratinocytes.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Wound Healing | 24 weeks post-treatment
  Proportion of RDEB wound sites with ≥50% healing from Baseline in treated versus untreated wounds
Pain Reduction | 24 weeks post-treatment
  Associated with wound dressing change assessed by the mean differences in scores of the Wong-Baker FACES scale between treated and untreated wounds

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Redwood City, California
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang JY, Marinkovich MP, Wiss K, McCarthy D, Truesdale A, Chiou AS, Eid E, McIntyre JK, Bailey I, Furukawa LK, Gorell ES, Harris N, Khosla RK, Peter Lorenz H, Lu Y, Nazaroff J, Grachev ID, Moore AJ. Prademagene zamikeracel for recessive dystrophic epidermolysis bullosa wounds (VIITAL): a two-centre, randomised, open-label, intrapatient-controlled phase 3 trial. Lancet. 2025 Jul 12;406(10499):163-173. doi: 10.1016/S0140-6736(25)00778-0. Epub 2025 Jun 23. PMID 40570869